CLINICAL TRIAL: NCT01167738
Title: A Randomized Phase II Study of Chemotherapy ± Metformin in Metastatic Pancreatic Cancer
Brief Title: Combination Chemotherapy With or Without Metformin Hydrochloride in Treating Patients With Metastatic Pancreatic Cancer
Acronym: PACT-17
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: concern of detrimental effect
Sponsor: IRCCS San Raffaele (Other)
Responsible Party: Principal Investigator, Michele Reni, MD, IRCCS San Raffaele
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000681691; PACT-17 (Other: IRCCS San Raffaele); 2010-020979-23 (EudraCT Number)
Record Dates: First submitted 2010-07-21; First posted 2010-07-22 (Estimated); Last update posted 2015-04-24 (Estimated); Status verified 2015-04

CONDITIONS: Pancreatic Cancer
Keywords: adenocarcinoma of the pancreas; stage IV pancreatic cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Capecitabine; Cisplatin; Epirubicin; Gemcitabine; Metformin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- PEXG regimen + metformin (Experimental): cisplatin and epirubicin at 30 mg/mq on days 1 and 15, capecitabine at 1250 mg/mq days 1-28, gemcitabine at 800 mg/mq on days 1 and 15, Metformin at 2 g days 1-28
  Interventions: Drug: capecitabine; Drug: cisplatin; Drug: epirubicin; Drug: gemcitabine; Drug: metformin
- PEXG regimen (Active Comparator): cisplatin and epirubicin at 30 mg/mQ on days 1 and 15, capecitabine at 1250 mg/mq days 1-28, gemcitabine at 800 mg/mq on days 1 and 15
  Interventions: Drug: capecitabine; Drug: cisplatin; Drug: epirubicin; Drug: gemcitabine

INTERVENTIONS:
Drug: capecitabine — 1250 mg/mq days 1-28 every 4 weeks
  Other Names: XELODA
Drug: cisplatin — 30 mg/mq on days 1 and 15 every 4 weeks
  Other Names: cisplatino TEVA
Drug: epirubicin — 30 mg/mq on days 1 and 15 every 4 weeks
  Other Names: farmorubicina
Drug: gemcitabine — 800 mg/mq on days 1 and 15 every 4 weeks
  Other Names: GEMZAR
Drug: metformin — 2 g days 1-28 every 4 weeks
  Other Names: glucophage
  Arms: PEXG regimen + metformin

SUMMARY:
RATIONALE: Drugs used in chemotherapy work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Giving more than one drug (combination chemotherapy) may kill more tumor cells. Metformin hydrochloride may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. It is not yet known if combination chemotherapy is more effective with or without metformin hydrochloride in treating patients with metastatic pancreatic cancer.

PURPOSE: This randomized phase II trial is studying giving cisplatin, epirubicin hydrochloride, capecitabine, and gemcitabine hydrochloride together with metformin hydrochloride to see how well it works compared to cisplatin, epirubicin hydrochloride, capecitabine, and gemcitabine hydrochloride alone in treating patients with metastatic pancreatic cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To assess the therapeutic activity of chemotherapy comprising cisplatin, epirubicin hydrochloride, capecitabine, and gemcitabine hydrochloride with versus without metformin hydrochloride in terms of 6-month progression-free survival in patients with metastatic pancreatic cancer.

Secondary

* To assess the overall survival of patients treated with this regimen.
* To assess the response rate in patients treated with this regimen.
* To assess the duration of response in patients treated with this regimen.
* To assess the toxicity in patients treated with this regimen.

OUTLINE: Patients are randomized to 1 of 2 treatment arms.

* Arm I: Patients receive cisplatin, epirubicin hydrochloride, and gemcitabine hydrochloride on days 1 and 15. Patients will also receive capecitabine and metformin hydrochloride on days 1-28. Treatment repeats every 4 weeks for up to 6 courses in the absence of disease progression or unacceptable toxicity.
* Arm II: Patients receive cisplatin, epirubicin hydrochloride, gemcitabine hydrochloride, and capecitabine as in arm I. Treatment repeats every 4 weeks for up to 6 courses in the absence of disease progression or unacceptable toxicity.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed pancreatic adenocarcinoma

  * Metastatic (stage IV) disease
* Measurable disease
* No symptomatic brain metastases

PATIENT CHARACTERISTICS:

* Karnofsky performance status 60-100%
* Not pregnant or nursing
* Adequate bone marrow, liver and kidney function
* No previous or concurrent malignancies at other sites except for surgically cured carcinoma in-situ of the cervix, basal cell or squamous cell carcinoma of the skin, or other neoplasms without evidence of disease within the past 5 years
* No multiple severe diseases which would compromise safety (i.e., cardiac failure, previous myocardial infarction within the past 4 months, cardiac arrhythmia, or history of psychiatric disabilities)
* No alcohol abuse

PRIOR CONCURRENT THERAPY:

* No prior chemotherapy or metformin
* No other concurrent experimental drugs

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2010-07; Primary Completion 2014-12 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Progression-free survival at 6 months | every 2 months
  CT scan

SECONDARY OUTCOMES:
Overall survival | every 14 days during therapy; every 3 months thereafter
  outpatient visit, phone interview
Response rate | every 2 months
  CT scan
Toxicity | every 2 weeks
  outpatient visit, laboratory findings

CONTACTS AND LOCATIONS:
Overall Officials: Michele Reni, MD, Principal Investigator — Istituto Scientifico H. San Raffaele
Locations (1):
- Istituto Scientifico H. San Raffaele, Milan, Italy